CLINICAL TRIAL: NCT00701467
Title: HRV Registry to Investigate Changes During the Time Before a Spontaneous Episode of Ventricular Tachyarrhythmia
Brief Title: Change in Heart Rate Variability Prior to Tachyarrhythmia in ICD Implanted Patients
Acronym: HRV
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Michael Glikson, Director , Davidai Arrhythmia Center, Leviev Heart Center, Sheba Medical Center
Other Study IDs: SHEBA-4743-07-MG-CTIL
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Ventricular Tachyarrhythmia
Keywords: ICD; ICD implanted patients
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation

SUMMARY:
To investigate changes in HRV during the time before a spontaneous episode of ventricular tachyarrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* S/P lexos VR/-T,DR/-T implantation
* Signed patient informed consent

Exclusion Criteria:

* CAF
* Life expectancy<6 months
* Impending heart transplant
* Persistent recurring tachycardia
* Rhythm disturbances that preclude a meaningful HRV analysis
* Participation in another study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ICD clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in RR interval recorded by ICD | within an hour before ventricular tachyarrythmia

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glikson, MD, Principal Investigator — SHEBA MC
Locations (1):
- Arrythmia Service Center, Ramat Gan, Israel